CLINICAL TRIAL: NCT04108429
Title: Expanding College Student Mental Health With Stress Management Mobile Technologies - Campus Wide Study
Brief Title: IntelliCare in College Students - Implementation (ICCS-I)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Emily G Lattie, Assistant Professor, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: K08MH112878-IET; K08MH112878 (NIH)
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Results first posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Depression; Anxiety
Keywords: Mental health; App; Mobile phone; Stress management
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Mobile self-help intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile self-help intervention (Experimental): Participants will have open access to the IntelliCare system.
  Interventions: Behavioral: IntelliCare for College Students

INTERVENTIONS:
Behavioral: IntelliCare for College Students — Participants will receive access to the IntelliCare system, which consists of apps with a variety of resources, including lessons and tools designed to teach skills for mood management. It is suggested that participants utilize the mobile phone tools every day

SUMMARY:
This study is a hybrid effectiveness-implementation trial of the smartphone student stress-management app IntelliCare for college students. This intervention will be tested with University of Illinois at Chicago (UIC) and Northern Illinois University (NIU) students. During the study, participants will complete measures of depressive and anxious symptoms, as well as measures of mental health literacy, within the app.

DETAILED DESCRIPTION:
In this study, students will be recruited to use the IntelliCare Hub app and encouraged to use it daily.The overall aim of this study is to pilot the program, evaluation metrics, implementation strategies, data collection and assessment procedures for a larger implementation trial. During the trial, participants will be prompted to complete the PHQ-8 and GAD-7 every week. At monthly intervals, participants will be prompted within the app to complete the Depression Literacy Questionnaire and Anxiety Literacy Questionnaire to measure mental health literacy, the Knowledge and Beliefs about Services scale to measure knowledge of campus mental health services, the Barriers to Mental Health Help-Seeking questionnaire to measure treatment barriers, and the Cognitive and Behavioral Response to Stress Scale to measure cognitive and behavioral coping skills. Counseling center utilization data will be extracted from the participating counseling centers' electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Participant is a student at the University of Illinois in Chicago or Northern Illinois University. *Participant owns a smartphone capable of running Android 7 (or higher) or iOS11 (or higher).
* Participant is 18 years of age or older

Exclusion Criteria:

*None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-02-05 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile Self-help Intervention
Started | 117
Completed | 117
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Mobile Self-help Intervention
Number analyzed (Participants) | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.27 (5.93)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 96
  Male | 17
  Other | 2
  Declined to respond | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 92
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 25
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 56
  More than one race | 15
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 117
Patient Health Questionnaire 8 (PHQ-8) depression score [Median (Full Range); unit: units on a scale] — The PHQ-8 measures depressive symptoms on a scale from 0-24 with higher score representing higher levels of depressive symptoms Population: Baseline PHQ and GAD data were collected within the app, and many participants did not complete the measures
  units on a scale
    number analyzed (Participants) | 73
    (all) | 10.5 [1 to 24]
Generalized Anxiety Disorder - 7-item questionnaire (GAD-7) score [Median (Full Range); unit: units on a scale] — The GAD-7 measures anxiety symptoms on a scale from 0-21 with higher score representing higher levels of anxiety symptoms Population: Baseline PHQ and GAD data were collected within the app, and many participants did not complete these measures
  units on a scale
    number analyzed (Participants) | 73
    (all) | 10 [0 to 21]

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire - 9 (PHQ-9) - Depression Severity Module
Description: The PHQ-9 measures degree of depression severity. Possible range of scores for the PHQ-9 is 0-27. Higher values represent a worse outcome.
  Specifically, scores of 0-4 indicate minimal or no depression; 5-9 is mild; 10-14 is moderate; 15-19 is moderately severe; and 20-27 is severe
Time Frame: Weekly symptom reports at Weeks 1, 2, 4, 6 and 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Self-help Intervention
Number analyzed (Participants) | 73
units on a scale
  Week 1 | 11.2 (15.5)
  Week 2 | 9.5 (15.4)
  Week 4 | 10.9 (17.5)
  Week 6 | 9.4 (17.7)
  Week 8 | 9.1 (15.4)
Statistical Analysis 1: Comparison: Mobile Self-help Intervention; generalized linear mixed model - this analysis accounts for repeated measures from each participant over the course of Weeks 1, 2, 4, 6 and 8; Test type: Superiority; p = .830, Mixed Models Analysis

2. Primary Outcome: Generalized Anxiety Disorder Scale - 7 (GAD-7)
Description: The GAD-7 is a self-administered 7 item instrument that uses some of the DSM-V criteria for GAD (General Anxiety Disorder) to identify probable cases of GAD along with measuring anxiety symptom severity. GAD-7 total score for the seven items ranges from 0 to 21. Higher values represent a worse outcome. Specifically, scores of 1-4 indicate minimal anxiety symptoms; 5-9 is mild anxiety symptoms; 10-14 is moderate anxiety symptoms; and 15-21 is severe anxiety symptoms.
Time Frame: Weekly symptom reports at Weeks 1, 2, 4, 6 and 8
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Self-help Intervention
Number analyzed (Participants) | 73
units on a scale
  Week 1 | 10.0 (7.7)
  Week 2 | 8.6 (10.6)
  Week 4 | 9.0 (6.9)
  Week 6 | 9.4 (14.2)
  Week 8 | 10.3 (10.9)
Statistical Analysis 1: Comparison: Mobile Self-help Intervention; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = .759, Mixed Models Analysis

3. Primary Outcome: Counseling Center Utilization Data (e.g. Counts of Individual Counseling Appointments)
Description: Counseling session utilization data were examined on a biweekly basis to determine if the introduction of the IntelliCare for College Students program impacts counseling center utilization. Counts of types of sessions (e.g. intake appointments, individual counseling appointments, crisis appointments) attended by students were examined over time to look at potential changes. These data were collected from the university in aggregate, thus, there are not participant-level data.
Time Frame: Biweekly session utilization from August 1, 2018 (start of pre-implementation data collection; prior to the implementation trial) to December 18, 2020 (end of implementation period)
Population: Data were collected from the counseling centers at both universities regarding how many appointments were scheduled each month from August 2018 to December 2020. For University A, August 2018 to January 2020 was labeled as the pre-implementation phase, and February 2020 to December 2020 was labeled as the implementation phase. For University B, August 2018 to July 2020 was labeled as the pre-implementation phase and August 2020 to December 2020 was labeled as the implementation phase.
Measure: Mean (Standard Deviation); unit: Appointments
Units Other Than Participants: Appointments
Groups:
- University A: Counseling Center Utilization at University A
- University B: Counseling Center Utilization at University B
Arm/Group | University A | University B
Number analyzed (Participants) | NA | NA
Number analyzed (Appointments) | 6580 | 18620
Appointments
  Intake - pre-implementation | 25.4 (18.2) | 117.1 (60.7)
  Intake - implementation | 9.7 (13.1) | 99.8 (37.4)
  Individual therapy - pre-implementation | 224.6 (138.3) | 531.5 (166.2)
  Individual therapy - implementation | 149.3 (85.1) | 442 (122.6)
  Crisis - pre-implementation | 3.3 (2.9) | 12.8 (10.1)
  Crisis - implementation | 1.7 (2.1) | 7 (4.2)
Statistical Analysis 1: Comparison: University A vs University B; Counseling center utilization data were examined using Simulation Modeling Analysis (SMA) for Time-Series data to determine if there were changes in utilization between the pre-implementation and implementation phases. SMA evaluates the statistical significance of between-phase changes in data streams and also accounts for the presence of autocorrelation (the non-independence of data points in time-series data streams); Test type: Superiority; p = .275, Simulation Modeling Analysis (SMA) for T

4. Primary Outcome: Average Number of Days of App Usage
Description: The mean number of days the app was used was drawn from the study app over the course of the study
Time Frame: Days of app use through study completion, up to 10 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mobile Self-help Intervention
Number analyzed (Participants) | 117
days | 6.29 (11)

5. Secondary Outcome: Anxiety Literacy Questionnaire
Description: This is a measure of mental health literacy, specifically about symptoms of anxiety. Participants respond "True" or "False" to statements about anxiety and the correct responses are tallied to create total score. The range of score is range of scores is 0-22 with higher scores indicating greater literacy.
Time Frame: Monthly questionnaire scores at baseline, one month and two months
Population: There was a substantial amount of missing data on this scale
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Self-help Intervention
Number analyzed (Participants) | 64
units on a scale
  Baseline | 14.4 (3.3)
  1 month | 15.6 (4.2)
  2 month | 14.1 (5.5)
Statistical Analysis 1: Comparison: Mobile Self-help Intervention; Test type: Superiority — generalized linear mixed model; p = .002, Mixed Models Analysis

6. Secondary Outcome: Depression Literacy Questionnaire
Description: This is a measure of mental health literacy, specifically about symptoms of depression. Participants respond "True" or "False" to statements about depression and the correct responses are tallied to create total score. The range of scores is 0-22 with higher scores indicating greater literacy.
Time Frame: Monthly questionnaire scores at baseline, one month and two months
Population: There was a substantial amount of missing data on this measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mobile Self-help Intervention
Number analyzed (Participants) | 42
units on a scale
  Baseline | 16.2 (2.9)
  1 month | 17.0 (3.5)
  2 month | 16.7 (2.9)
Statistical Analysis 1: Comparison: Mobile Self-help Intervention; generalized linear mixed model; Test type: Superiority; p = .489, Mixed Models Analysis

7. Secondary Outcome: Cognitive and Behavioral Response to Stress Scale (CB-RSS)
Description: The CB-RSS is a 9 item measure of the frequency and perceived helpfulness of cognitive and behavioral coping skills. There are 4 subscales representing "Cognitive frequency" "Cognitive helpfulness" "Behavioral frequency" and "Behavioral helpfulness." Participants respond to the frequency items on a scale of 0 = Never to 6 = Always and to the helpfulness items on a scale of 0 = Not at all helpful to 6 = Extremely helpful. The scores range from 0-24 on the Cognitive subscales and from 0-30 on the Behavioral subscales. Higher values represent a better outcome.
Time Frame: Monthly questionnaire scores at baseline, one month and two months
Population: There was a substantial amount of missing data on this scale
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Self-help Intervention
Number analyzed (Participants) | 36
score on a scale
  CB-RSS Cognitive Frequency Baseline | 9.9 (5.1)
  CB-RSS Cognitive Frequency 1 month | 11.2 (6.4)
  CB-RSS Cognitive Frequency 2 month | 8.02 (5.8)
  CB-RSS Cognitive Usefulness Baseline | 9.5 (5.7)
  CB-RSS Cognitive Usefulness 1 month | 9.7 (6.8)
  CB-RSS Cognitive Usefulness 2 month | 7.3 (8.7)
  CB-RSS Behavioral Frequency Baseline | 11.6 (4.9)
  CB-RSS Behavioral Frequency 1 month | 11.0 (8.4)
  CB-RSS Behavioral Frequency 2 month | 8.5 (5.4)
  CB-RSS Behavioral Usefulness Baseline | 14.9 (6.8)
  CB-RSS Behavioral Usefulness 1 month | 17.0 (11.0)
  CB-RSS Behavioral Usefulness 2 month | 8.4 (8.6)
Statistical Analysis 1: Comparison: Mobile Self-help Intervention; generalized linear mixed model; Test type: Superiority; p = .001, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | Mobile Self-help Intervention
All-Cause Mortality (participants affected / at risk) | 0/117
Serious Adverse Events (participants affected / at risk) | 0/117
Other Adverse Events (participants affected / at risk) | 0/117

LIMITATIONS AND CAVEATS:
Due to COVID-19-related changes and ongoing uncertainty surrounding operations on the university campuses with which we partnered, many of the program implementation plans were unable to be enacted. Due to the in-app nature of assessments, there was a high degree of data missingness on the mental health symptom data and the intervention target data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT04108429/Prot_SAP_ICF_000.pdf